CLINICAL TRIAL: NCT02372474
Title: "It is a Real" The First Baby Of Autologous Stem Cell Therapy in Premature Ovarian Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Edessy Mahmoud, Professor, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M Edessy
Record Dates: First submitted 2015-01-12; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Premature Ovarian Failure
Keywords: POF; ESS; stem cell therapy
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cell therapy in POF (Experimental): POF cases were evaluated hormonally, HP and IH using ESS. Autologous MSC were prepared and laparoscopically transplanted.
  Interventions: Biological: Stem cell

INTERVENTIONS:
Biological: Stem cell — Out of 112 high risk patients for POF diagnosis was established in 10 cases. Endometrial fractional biopsy was taken, stained with H&E stain and by Immunohistochemical (IH) staining by stem cell marker OCT4. IH expression of stem cell was evaluated before and after transplantation according to Edessy Stem Cell Scoring (ESS). After laparoscopic injection of stem cell sample in the ovaries, participants were followed up monthly for a period of one year by hormonal (FSH, LH and E2), clinical (resuming menstruation and pregnancy), US (folliculometry), histopathological (HP), and IH expression of stem cell (stem cell positivity and scoring according to ESS).
  Other Names: - Edessy Stem cell Score.; - Laparoscopic stem cell transplantation.; - Hormonal Analysis; - Ultrasonic evaluation

SUMMARY:
The purpose of this work is to evaluate the therapeutic potential of Autologous Mesenchymal sc (MSC) therapy in women suffering from POF.

DETAILED DESCRIPTION:
Stem cells (sc) are the foundation cells for every organ, tissue and cell in the body. They are self sustaining and can replicate themselves for long periods of time. They have the remarkable potential to develop in many different cell types in the body. Premature ovarian failure (POF) is the loss of ovarian function in women less than 40 years. It is associated with sex steroid deficiency, amenorrhea, infertility, and elevated serum gonadotropins. This work aimed to evaluate the therapeutic potential of Autologous Mesenchymal sc (MSC) transplantation in women suffering from POF. Out of 112 high risk patients for POF, 10 cases were diagnosed as POF. The ten POF patients were scheduled for MSC transplantation at Al- Azhar University Hospitals. MSC preparation from the bone marrow of the iliac crest was laparoscopically injected in the ovaries. Endometrial fractional biopsy is histopathologically (HP) and Immunohistochemically (IH) stained and evaluated according to Edessy stem cells score (ESS) (1).

ELIGIBILITY:
Inclusion Criteria:

* Post-menarche female less than 40 years old.
* Normal karyotyping female.
* Primary ovarian failure females
* Follicle-stimulating hormone (FSH) more than or equal to 20 IU/L.
* Agree to sign the designed consent for the study.

Exclusion Criteria:

* Autoimmune diseases.
* Breast cancer, ovarian cancer.
* Hypersensitivity to any Gonadotropin-releasing hormone (GnRH) analogs.
* Those with major medical problems such as malignancy, hepatitis, etc.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of cases go through menstruation, pregnancy and labour after stem cell transplantation in POF. | 128 weeks
  Cases underwent sc transplantation were followed up for occurrence of menstruation and pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Edessy, Professor, Principal Investigator — Al-Azhar University; Hala N Hosni, Professor, Study Chair — Cairo University; Yousef Shdy, MD, Study Chair — Al-Azhar University; Syed Bkry, MD, Study Chair — Al-Azhar University; Medhat Kamel, Msc, Study Chair — Al-Azhar University
Locations (1):
- Al Azhar University, Cairo, Cairo Governorate, Egypt